CLINICAL TRIAL: NCT01589172
Title: Evaluating the Use of Thromboelastography to Diagnose and Monitor Coagulopathy Associated With Pediatric Traumatic Brain Injury
Brief Title: Evaluating the Use of Thromboelastography to Diagnose Coagulopathy After Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Sponsor
Other Study IDs: 120296
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Traumatic Brain Injury; Coagulation Disorder
MeSH Terms: conditions — Brain Injuries, Traumatic; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric Brain Trauma Patients

SUMMARY:
The investigators will obtain thromboelastography (TEG) on pediatric patients admitted to the Rady Children's Hospital ICU after traumatic brain injury on admission to our ICU and after 24 hours of care. The investigators hypothesize that TEG will identify abnormalities of coagulation that are not identified by traditional coagulation studies, i.e. prothrombin time (PT), activated partial thromboplastin time (aPTT), and international normalized ratio (INR).

ELIGIBILITY:
Inclusion Criteria:

* less than 15 years of age
* evidence of intracranial bleed on CT scan or GCS <12

Exclusion Criteria:

* No intracranial hemorrhage or
* GCS 13 - 15

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Trauma patients admitted to the Rady Children's Hospital Pediatric Intensivse Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2012-11-30 (Actual); Study Completion 2012-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David K Shellington, MD, Principal Investigator — University of California, San Diego
Locations (1):
- Rady Children's Hospital, San Diego, California, United States